CLINICAL TRIAL: NCT04698239
Title: Clinical Evaluation of the Safety and Benefits of the Milesman 445 nm Blue Laser on Inflammatory Acne Lesions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaias Salud (Network)
Collaborators: Gaias Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MILESMAN-ACNE
Record Dates: First submitted 2020-10-06; First posted 2021-01-06 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris; LASER
Keywords: LASER; ACNÉ; MILESMAN
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser application ( BEFORE/AFTER) (Experimental): All patients will receive a maximum of 13 laser pulses in each lesion. We are going to make a comparison of the before and after the treatment, it is the patient himself who checks himself.
  The number of lesions will be counted before treatment and after treatment(72-hour and 1-week ) . Adverse reactions will be collected at several visits as well, during the 2 weeks that the patient is included in the study.
  Interventions: Device: LASER MILESMAN 445 NM

INTERVENTIONS:
Device: LASER MILESMAN 445 NM — Laser application

SUMMARY:
Acne treatment by laser or other light devices is a currently accepted procedure. It allows faster resolution of injuries, with fewer side effects and greater patient satisfaction.

The mechanism of action of the Milesman Blauman laser is based on diode laser technology that produces pulses of blue light with a wavelength of 445 nanometers, in the blue and visible spectrum. It combines the precision of laser technology by focusing energy on diseased areas.

DETAILED DESCRIPTION:
Introduction / Justification Acne vulgaris (AV) is a polygenic multifactorial disease of the pilosebaceous units, which leads to the formation of both non-inflammatory lesions (comedones) and inflammatory lesions (papules, pustules, nodules and cysts), which affects approximately 85% of the population .

Acne treatment by laser or other light devices is a currently accepted procedure. It allows faster resolution of injuries, with fewer side effects and greater patient satisfaction.

The mechanism of action of the Milesman Blauman laser is based on diode laser technology that produces pulses of blue light with a wavelength of 445 nanometers, in the blue and visible spectrum. It combines the precision of laser technology by focusing energy on diseased areas.

The MILESMAN Laser has been on the market for over two years and has been used for cosmetic purposes and has proven to be safe during that time on the market.

MAIN GOAL The main objective of this study is to describe the efficacy and safety of the device (Milesman Laser) as a treatment for inflammatory acne lesions (papules and pustules). To do this, we will measure the evolution of the number of injuries of this type on the patient, before and after the application of the laser.

EXPLORATORY OBJECTIVES

Additionally, the study will have the following objectives:

* Exploratory assessment of the change in acne classification on the EGAE scale (grade 1 - 4) after laser application.
* Evaluate the adverse effects derived after the laser application.
* Evaluate the degree of patient satisfaction after the laser application. STUDY DESIGN Open, prospective, interventional, single-arm, quasi-experimental analytical study of before and after.

This type of design is based on the measurement and comparison of the response variable before and after the subject's exposure to the experimental intervention. It is a national, single-center study.

SAMPLE SIZE According to the objective of the study, we plan to get at least 25 patients. In this study we define sample as the entire area to be treated on the face, that is, we will obtain 25 samples.

STUDY PERIOD The duration of the study will be 3 months from the inclusion of the first patient. The duration of the patient in the study is 14 days.

DESCRIPTION OF THE INTERVENTION The Milesman laser has a handpiece, which allows each injury to be targeted via an indicator light and the person handling it will trigger the shot via a foot pedal. A maximum of 10 shots will be made on each acne injury, depending on the size and type of injury. Finally, 2-3 shots will be taken to photocoagulate the follicle walls and thus prevent the lesion from recurring or becoming infected again.

The laser will be applied to all inflammatory facial injuries in a single session, it is estimated that the duration of the session is about 20 minutes, depending on the number of injuries

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 50 years old
* Diagnosis of mild to moderate acne on the face
* They must have 10 - 50 inflammatory lesions (papules and pustules) on the face
* In general good health

Exclusion Criteria:

* Allergies or light sensitivities.
* Severe acne or pre-existing dermatological facial condition
* Presence of cysts on the face
* More than one nodule on the face
* Having an uncontrolled disease or an immunodeficient disorder.
* Being pregnant or lactating
* Oral and / or topical antibiotic treatment in the last 2 weeks.
* Current treatment with hormonal contraceptives.
* Impossibility of avoiding excessive sun exposure and any light treatment or any similar pro-fessional or aesthetic procedure during the 15 days before and 15 days after treatment.
* Previous history of poorly healed wounds, keloid formation, or bleeding disorders
* Process of active or historical infection of herpes simplex.
* Extreme sensitivity to hydroquinone or other bleaching agents.
* Personal or family history of melanoma.
* Dysplastic nevus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
How many lesions treated have disappeared | 1 week
  Number of lesions before laser vs. number of lesions after laser(72 h and 1 week ).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by MedRA | 2 weeks
  The number of related adverse reactions is collected and cataloged.

CONTACTS AND LOCATIONS:
Locations (1):
- GAIAS RESEARCH,C/PINTOR XAIME QUESADA Nº3, Santiago de Compostela, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: No